CLINICAL TRIAL: NCT02416388
Title: Phase II/III Randomized Study to Improve Overall Survival in 18 to 60 Year-old Patients, Comparing Daunorubicin Versus High Dose Idarubicin Induction Regimens, High Dose Versus Intermediate Dose Cytarabine Consolidation Regimens, and Standard Versus Mycophenolate Mofetil Prophylaxis of Graft Versus Host Disease in Allografted Patients in First CR : a Backbone InterGroup-1 Trial
Brief Title: Study to Improve OS in 18 to 60 Year-old Patients, Comparing Daunorubicin Versus High Dose Idarubicin Induction Regimens, High Dose Versus Intermediate Dose Cytarabine Consolidation Regimens, and Standard Versus MMF Prophylaxis of GvHD in Allografted Patients in First CR
Acronym: BIG-1
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC-2010-03
Record Dates: First submitted 2015-04-07; First posted 2015-04-15 (Estimated); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Idarubicin; Daunorubicin; Cyclosporine; Methotrexate; Mycophenolic Acid; vosaroxin; Dexamethasone; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (14):
- R1-IDA (Experimental): Idarubicin
  Interventions: Drug: Idarubicin
- R1-DAUNO (Active Comparator): Daunorubicin
  Interventions: Drug: Daunorubicin
- R2-HDAC (Active Comparator): High dose cytarabine
  Interventions: Drug: HD Cytarabine
- R2-IDAC (Experimental): Intermediate dose cytarabine
  Interventions: Drug: ID cytarabine
- R3-MAC-MTX (Active Comparator): Methotrexate and mycophenolic acid
  Interventions: Drug: Methotrexate; Drug: Mycophenolic acid (MPA)
- R3-MAC-MPA (Experimental): Cyclosporine and mycophenolic acid
  Interventions: Drug: Cyclosporine; Drug: Mycophenolic acid (MPA)
- R3-RIC-CICLO (Active Comparator): Cyclosporine
  Interventions: Drug: Cyclosporine
- R3-RIC-MPA (Experimental): Cyclosporine and mycophenolic acid
  Interventions: Drug: Cyclosporine; Drug: Mycophenolic acid (MPA)
- R4-VOS-IDAC (Experimental): Intermediate dose cytarabine and vosaroxin
  Interventions: Drug: vosaroxin; Drug: ID cytarabine
- R4-IDAC (without VOS) (Active Comparator): Intermediate dose cytarabine alone
  Interventions: Drug: ID cytarabine
- R4-DEX-HDAC (Experimental): High dose cytarabine and dexamethasone
  Interventions: Drug: HD Cytarabine; Drug: Dexamethasone
- R4-HDAC (without DEX) (Active Comparator): High dose cytarabine alone
  Interventions: Drug: HD Cytarabine
- R4-VEN-IDAC (Experimental): Intermediate dose cytarabine and venetoclax
  Interventions: Drug: ID cytarabine; Drug: Venetoclax
- R4-IDAC (without VEN) (Active Comparator): Intermediate dose cytarabine alone
  Interventions: Drug: ID cytarabine

INTERVENTIONS:
Drug: Idarubicin — Induction chemotherapy :
  Idarubicin 9mg/m² /day, from D1 to D5 (IV, 30min)
  + cytarabine 200mg/m²/day from D1 to D7 (IV 24 h)
  Bone marrow aspirate on D15 : if medullary blasts rate < 5% → G-CSF (5 μg/kg/day) until hematopoietic recovery (PNN ≥ 1 G/L).
  Arms: R1-IDA
Drug: Daunorubicin — Induction chemotherapy :
  Daunorubicin 90mg/m²/day, from D1 to D3 (IV, 30min)
  + cytarabine 200mg/m² /day from D1 to D7 (IV 24 h)
  Bone marrow aspirate on D15 : if medullary blasts rate < 5% → G-CSF (5 μg/kg/day) until hematopoietic recovery (PNN ≥ 1 G/L).
  Arms: R1-DAUNO
Drug: HD Cytarabine — Consolidation chemotherapy course (s) :
  -High dose cytarabine: 3g/m² /12h on D1, D3 and D5
  For all patients, G-CSF (5 μg/kg/day) : SC or IV (30 min) from D8 until hematopoietic recovery (PNN ≥ 1 G/L)
  Up to 3 consolidation courses, depending on the patient AML risk group
  Arms: R2-HDAC; R4-DEX-HDAC; R4-HDAC (without DEX)
Drug: Cyclosporine — GvHD prophylaxis post allogeneic SCT :
  -Cyclosporine : 3 mg/kg /day from D-1 (IV) or 6 mg/kg/day from D-3 (PO). Not to be stopped before D100
  Arms: R3-MAC-MPA; R3-RIC-CICLO; R3-RIC-MPA
Drug: Methotrexate — GvHD prophylaxis post allogeneic SCT :
  -15 mg/m² on D+1 then 10 mg/m² on D+3, D+6 and D+11
  Arms: R3-MAC-MTX
Drug: Mycophenolic acid (MPA) — GvHD prophylaxis post allogeneic SCT :
  * 720 mg BID from D0 to D+28 for HLA-identical siblings
  * 720 mg BID from D0 to D+45 for 10/10 HLA allele-matched unrelated donors
  Arms: R3-MAC-MPA; R3-MAC-MTX; R3-RIC-MPA
Drug: vosaroxin — Consolidation chemotherapy course (s) :
  -70 mg/m² on D1 and D4
  Arms: R4-VOS-IDAC
Drug: ID cytarabine — Consolidation chemotherapy course (s) :
  -Intermediate dose cytarabine: 1.5g/m² /12h on D1, D3 and D5
  For all patients, G-CSF (5 μg/kg/day) : SC or IV (30 min) from D8 until hematopoietic recovery (PNN ≥ 1 G/L)
  Up to 3 consolidation courses, depending on the patient AML risk group
  Arms: R2-IDAC; R4-IDAC (without VEN); R4-IDAC (without VOS); R4-VEN-IDAC; R4-VOS-IDAC
Drug: Dexamethasone — Consolidation chemotherapy course (s) :
  -10 mg/12h on D1, D3 and D5
  Arms: R4-DEX-HDAC
Drug: Venetoclax — Consolidation chemotherapy course (s) :
  Once RP2D has been determined from the results of the dose selection phase (phase 1), the optimal dose level retained for randomized phase 2 will be one of the following:
  * 100 mg/d on D1 to D8 (selection phase dose level 1)
  * or 200 mg/d on D1 to D8 (selection phase dose level 2)
  * or 400 mg/d on D1 to D8 (selection phase dose level 3)
  * or 400 mg/d on D1 to D14 (selection phase dose level 4)
  Arms: R4-VEN-IDAC

SUMMARY:
This open label, multicenter phase II/III study with multiple randomization phases at differents stages of AML treatment (induction, consolidation and HSCT where applicable) is designed to improve OS in younger (18 to 60 year-old) patients, with AML risk-adapted patient strategies. Within the intermediate risk AML group, optimal GvHD prophylaxis following allogeneic SCT in first CR, after either myeloablative (MAC) or reduced intensity (RIC) conditioning, will also be evaluated. With an adaptative design, this clinical trial could test up to 3 novel AML agents of interest.

ELIGIBILITY:
Inclusion Criteria (at diagnosis) :

1. Age ≥ 18 years and < 61 years
2. With a newly diagnosed de novo or secondary type AML (post myelodysplastic syndrome MDS or therapy-related AML)
3. No prior treatment for neither AML (with the exception of hydroxyurea), nor MDS (with the exception of EPO)
4. ECOG performance status ≤ 3
5. Absence of severe uncontrolled infection
6. No cardiac contraindications for the use of anthracyclines : decompensated or uncontrolled heart failure, recent myocardial infarction, current signs of cardiac impairment, uncontrolled arrhythmias, LVEF (left ventricular ejection fraction) < 50%
7. Total bilirubin ≤ 2 x upper limit of normal (UNL), ASAT(SGOT) and ALAT (SGPT) ≤ 2.5 X UNL, creatinine < 150 µmol/l, unless AML-related out of range values
8. Genetic mutation testing of the FLT3 (FLT3-ITD ou FLT3-TKD) gene, performed in local or central laboratory
9. Use of appropriate methods of contraception:

   * for patients treated with Midostaurin:

     * women of childbearing potential should use appropriate methods of contaception throughout treatment, and for 5 months post cessation of treatment
     * men will need to use condoms during intercourse throughout treatment, and for 5 months post cessation of treatment with Midostaurin
10. Patients who are covered by or beneficiaries of a social security system (Social Security or Universal Medical Coverage)
11. Patients who have read and understood the information sheet and signed the informed consent form

Exclusion criteria (at diagnosis) :

1.Patients with acute promyelocytic leukemia (APL), as confirmed either by t(15;17) or by the presence of PML-RARA fusion transcripts 2.Patients with core binding factor (CBF) AML, as confirmed either by t(8;21), t(16,16) or inv(16), or by fusion transcripts resulting from these cytogenetic abnormalities (RUNX1-RUNX1T1, CBFB-MYH11).

3.Patients with secondary AML arising from myeloproliferative disorders previously known according to the 2008 WHO classification 4.Patients with Ph1+ AML or previous Ph1+ disorder (chronic myelogenous leukemia) 5.Severe psychiatric or organic disorder, supposed to be independent from AML, that would contraindicate treatment, including allogeneic HSCT 6.No psychological, familial, social, or geographic reason that would compromise clinical follow up 7.History of uncontrolled cancer for the last 2 years, with the exception of basal cell carcinoma or carcinoma in situ of the cervix 8.Uncontrolled severe infection 9.Patients with positive serology for HIV-1 and -2, or HTLV -1 and -2, or active hepatitis virus B or C infection 10.Pregnant or lactating women 11.Legal incapacity (patients under tutorship, curatorship or judicial protection)

------------------------------------------

For randomization R4-VOS (post-induction/salvage) :

Inclusion criteria

1. Patients enrolled in the BIG-1 trial at diagnosis
2. Patient presenting with AML in first CR or CRp/CRi after induction or one cycle of salvage therapy (confirmed in the 15 days preceding R4-VOS)
3. Favorable or intermediate risk AML patients, as stratified with BIG-1 prognostic classification
4. Patients randomized to R2-IDAC arm (intermediate dose cytarabine)
5. ECOG performance status ≤ 2
6. Left ventricular ejection fraction (LVEF) at least 40% by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO)
7. Local clinical laboratory values as follows:

   o Serum creatinine ≤ 2.0 mg/dL

   o Total bilirubin ≤ 1.5 X the upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) ≤ 2.5 X ULN
   * Alanine aminotransferase (ALT) ≤ 2.5 X ULN
8. Signed written informed consent for vosaroxin study (R4-VOS)
9. Women of childbearing potential must have a negative pregnancy test within 8 days before randomization R4-VOS and commit to the use of effective contraception during the period of treatment and up to 36 days after vosaroxin has been stopped. Men must use effective contraception during the treatment period and up to 96 days after vosaroxin has been stopped.

Exclusion criteria

1.Patients classified in the unfavorable risk group according to the BIG-1 protocol classification 2.Complete remission is not attained (CR, CRp/CRi) after induction and/or salvage therapy 3.Positive pregnancy test 4.Severe uncontrolled infection such as sepsis, or multiple organ dysfunction syndrome, uncontrolled fever 5.Documented uncontrolled fungal infection (positive blood test and cultures) 6.History of myocardial infarction, unstable angina, cerebrovascular accident (CVA) or transient ischemic attack (TIA) in the 3 months before randomization 7.Patient under hemodialysis (HD) or peritoneal dialysis (PD)

------------------------------------------

For randomization R4-DEX (post-induction/salvage) :

Inclusion criteria

1. Patients enrolled in the BIG-1 trial at diagnosis
2. Patient presenting with AML in first CR or CRp/CRi after induction or one cycle of salvage therapy (confirmed in the 15 days preceding R4-DEX)
3. Favorable or intermediate risk AML patients, as stratified with BIG-1 prognostic classification
4. ECOG performance status ≤ 2
5. Local clinical laboratory values as follows:

   * Serum creatinine ≤ 150 µmol/L
   * Total bilirubin ≤ 1.5 X the upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) ≤ 2.5 X ULN
   * Alanine aminotransferase (ALT) ≤ 2.5 X ULN
6. Signed written informed consent for dexamethasone study (R4-DEX)

Exclusion criteria

1.Severe uncontrolled infection such as sepsis, or multiple organ dysfunction syndrome, uncontrolled fever 2.Documented uncontrolled fungal infection (positive blood test and cultures 3.History of myocardial infarction, unstable angina, cerebrovascular accident (CVA) or transient ischemic attack (TIA) in the 3 months before randomization 4.Patient under hemodialysis (HD) or peritoneal dialysis (PD)

--------------------------------------

For randomization R4-VEN (post-induction/salvage) :

Inclusion criteria

1. Age 18 - 60 years at inclusion in BIG-1 protocol
2. diagnosis of AML according to WHO classification de novo or secondary to myelodysplastic syndrome (myelodysplastic syndrome must not have been treated except by ESA, Lenalidomide or non-chemotherapy) or therapy-related AML
3. Patients included in the BIG-1 protocol
4. Patients in first CR or CRp/CRi following 1 or 2 courses of induction chemotherapy according to BIG-1 protocol and who are planned to receive consolidation.
5. Patients stratified within the favorable and intermediate risk groups as defined by BIG-1 protocol
6. ECOG performance status ≤ 2
7. Left ventricular ejection fraction (LVEF) at least 40% by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO)
8. Creatinine clearance ≥ 30 ml/min (calculated by the usual method of each institution), total bilirubin ≤ 1.5 times the ULN; ASAT and ALAT ≤ times the upper limit of normal (ULN)
9. Absence of uncontrolled infection
10. Women of childbearing potential must agree to use effective contraception without interruption throughout the study and for a further 3 months after the end of treatment
11. Written signed informed consent

Exclusion criteria

1.AML stratified in the unfavorable BIG-1 risk-group. 2.Diagnosis of Acute Promyelocytic Leukemia or CBF AML (ie. AML with t(8;21), t(16,16) or inv(16), or their molecular equivalents RUNX1-RUNX1T1 and CBFB-MYH11) 3.AML secondary to prior myeloproliferative disorder according to WHO classification (2008) and Philadelphia chromosome-positive AML (Ph1+) 4.Absence of CR/CRp/CRi after a maximum of two chemotherapy cycles 5.Severe medical or mental condition precluding the administration of protocol treatments 6.Prior history of cancer unless controlled for at least 2 years and except for basocellular cutaneous cancers and in situ cervix cancers 7.Positive pregnancy test 8.Breast feeding 9.Uncontrolled infection such as sepsis, or multiple organ dysfunction syndrome, uncontrolled fever 10.Documented uncontrolled fungal infection (positive blood test and cultures) 11.Prior venetoclax exposure 12.Known HBV with detectable viral load 13.Known HIV positive patients 14.Known hypersensitivity to any of the study medication 15.History of myocardial infarction, unstable angina, cerebrovascular accident (CVA) or transient ischemic attack (TIA) in the 3 months before randomization 16.Patient under hemodialysis (HD) or peritoneal dialysis (PD) 17.Concomitant treatment with cytochrome CYP3A4 inhibitor which cannot be stopped during venetoclax administration ONLY FOR PHASE 1 18.During the phase 2, for patients randomized in the IDAC + Venetoclax arm, if concomitant treatment with cytochrome CYP3A4 inhibitor cannot be stopped, a dose reduction of 70% of venetoclax must be apply

--------------------------------------

For randomization R3 (before AlloHSCT):

Inclusion criteria

1. Patients enrolled in the BIG-1 trial at diagnosis
2. Patient presenting with AML in first CR or CRp/CRi treated in the BIG-1 trial and classified in the intermediate risk group, namely:

   * either initially favorable but poor molecular responders for NPM1 MRD: NPM1 mutation, without FLT3-ITD mutation or with an FLT3-ITD ratio < 0.50 and MRD2 positive blood (decrease of less than 4 log from baseline at diagnosis)).
   * Or initially favorable but requiring two cycles of chemotherapy (a salvage therapy) to obtain the first CR/CRp/CRi
   * Or other immediate intermediaries
3. No metastatic or progressive cancer, with the exception of basal cell skin carcinoma and cervical carcinoma in situ
4. Patients with general condition preserved (ECOG ≤ 3) and with no uncontrolled severe infection
5. Women of childbearing age must make use of effective contraception
6. Patients who are covered by or beneficiaries of a social security system (Social Security or Universal Medical Coverage).
7. Patients who have read and understood the information sheet and signed the informed consent form

Exclusion criteria

1. Complete remission is not obtained (CR, CRp/CRi) after induction and/or salvage therapy
2. Patient presenting with AML in first CR or CRp/CRi treated in the BIG-1 trial and classified either in the favorable risk group or the unfavorable risk group
3. Patients with a severe organ or psychiatric pathology, presumed to be independent of AML and contraindicating the allograft
4. Patients who, for family, social or geographic reasons, do not wish to be regularly monitored via consultation
5. Uncontrolled severe infection at the time of inclusion
6. Serology positive for HIV 1 or 2 or HTLV 1 or 2, or active HBV or HCV viral infection
7. Pregnant women (beta-HCG positive) or currently breastfeeding
8. Adult patient who is incapacitated, under wardship, legal guardianship, or under the protection of the courts
9. Patients under State Medical Assistance (AME)

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3100 (Estimated)
Dates: Start 2015-01; Primary Completion 2025-07 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years
  For randomizations R1 (idarubicine vs daunorubicine) and R2 (HDAC vs IDAC)
Cumulative incidence (CI) of acute Graft versus Host Disease (GvHD) of grade II to IV | 100 days
  For randomization R3 : GvHD prophylaxis study
Disease free survival | 18 months
  For randomizations R4

CONTACTS AND LOCATIONS:
Locations (56):
- France (56):
  - CH Amiens Hôpital Sud, Amiens
  - CHU Angers, Angers
  - CH Victor Dupouy, Argenteuil
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Hôpital Jean Minjoz, Besançon
  - CH Beziers, Béziers
  - Hôpital Avicenne, Bobigny
  - CH Bordeaux, Bordeaux
  - Hôpital du Dr Duchenne, Boulogne-sur-Mer
  - Hôpital Morvan, Brest
  - CH Caen, Caen
  - Clinique du parc, Castelnau-le-Lez
  - Centre Hospitalier René Dubos, Cergy-Pontoise
  - HIA Percy, Clamart
  - CHU Estaing, Clermont-Ferrand
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Hôpital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CH Dunkerque, Dunkirk
  - Hôpital Michallon, Grenoble
  - CH Versailles, Le Chesnay
  - CH Lens, Lens
  - CHRU de Lille, Hôpital Huriez, Lille
  - Hôpital St Vincent de Paul, Lille
  - CHU de Limoges, Limoges
  - Centre Leon Berard (CLB), Lyon
  - CH Lyon Sud, Lyon
  - Marseille La Conception, Marseille
  - Institut Paoli Calmettes, Marseille
  - CH Meaux, Meaux
  - CHR Metz Thionville_Hôpital de Mercy, Metz
  - Hôpital Saint Eloi, Montpellier
  - CH Mulhouse, Mulhouse
  - CH Hôtel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU Nice, Nice
  - CHRU de Nîmes, Nîmes
  - Hôpital Cochin, Paris
  - Hôpital La Pitié Salpêtrière, Paris
  - Hôpital Necker Enfants Malades, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital St Louis, Paris
  - Centre Hospitalier Saint Jean, Perpignan
  - CHU de Poitiers, Poitiers
  - Hôpital Robert Debré, Reims
  - CH Pontchaillou, Rennes
  - Hopital Victor Provo, Roubaix
  - Centre Henri Becquerel, Rouen
  - Hôpital René Huguenin, Saint-Cloud
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Hôpital Hautepierre, Strasbourg
  - IUCT Toulouse, Toulouse
  - CHU Bretonneau, Tours
  - CH Valenciennes, Valenciennes
  - Hôpitaux de Brabois_CHU Nancy, Vandœuvre-lès-Nancy
  - Institut de Cancérologie Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Hunault M, Pautas C, Bertoli S, Dumas PY, Raffoux E, Hospital MA, Marchand T, Heiblig M, Chantepie S, Carre M, Peterlin P, Gallego-Hernanz MP, Lemasle E, Guieze R, Simand C, Turlure P, Huynh A, Leguay T, Devillier R, Quoc SN, Duployez N, Luquet I, Penther D, Celli-Lebras K, Mineur A, Raus N, Gardin C, Socie G, Cahn JY, Ifrah N, Vey N, de Latour RP, Delabesse E, Preudhomme C, Hamel JF, Pigneux A, Recher C, Dombret H. Intermediate-Dose Cytarabine as Postinduction AML Therapy. NEJM Evid. 2025 Jul;4(7):EVIDoa2400326. doi: 10.1056/EVIDoa2400326. Epub 2025 Jun 24. PMID 40552969